CLINICAL TRIAL: NCT02875873
Title: Balanced Solution Versus Saline in Intensive Care Study
Acronym: BaSICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: basics001
Record Dates: First submitted 2016-08-15; First posted 2016-08-23 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Critical Illness; Acute Kidney Injury
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury | interventions — Plasma-lyte 148; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Plasma-Lyte, Slow Infusion (Experimental): Plasma-Lyte will be used for fluid expansion and maintenance whenever needed and when there is no contraindication either for Plasma-Lyte or normal saline. Whenever fluid expansion is deemed necessary by the attending physician, infusion speed will be set at 333 mL/h.
  Interventions: Drug: Plasma-Lyte; Other: Slow infusion speed
- Plasma-Lyte, Fast Infusion (Experimental): Plasma-Lyte will be used for fluid expansion and maintenance whenever needed and when there is no contraindication either for Plasma-Lyte or normal saline. Whenever fluid expansion is deemed necessary by the attending physician, infusion speed will be set at 999 mL/h.
  Interventions: Drug: Plasma-Lyte; Other: Fast Infusion Speed
- Saline 0.9%, Slow Infusion (Experimental): Saline 0.9% will be used for fluid expansion and maintenance whenever needed and when there is no contraindication either for Plasma-Lyte or normal saline. Whenever fluid expansion is deemed necessary by the attending physician, infusion speed will be set at 333 mL/h.
  Interventions: Drug: Saline 0.9%; Other: Slow infusion speed
- Saline 0.9%, Fast Infusion (Experimental): Saline 0.9% will be used for fluid expansion and maintenance whenever needed and when there is no contraindication either for Plasma-Lyte or normal saline. Whenever fluid expansion is deemed necessary by the attending physician, infusion speed will be set at 999 mL/h.
  Interventions: Drug: Saline 0.9%; Other: Fast Infusion Speed

INTERVENTIONS:
Drug: Plasma-Lyte — Plasma-Lyte will be used for fluid expansion and maintenance
  Arms: Plasma-Lyte, Fast Infusion; Plasma-Lyte, Slow Infusion
Drug: Saline 0.9% — Saline 0.9% will be used for fluid expansion and maintenance
  Other Names: Normal Saline
  Arms: Saline 0.9%, Fast Infusion; Saline 0.9%, Slow Infusion
Other: Slow infusion speed — Whenever fluid expansion is deemed necessary by the attending physician, infusion speed will be set at 333 mL/h. NOTE: This intervention will not be blinded.
  Arms: Plasma-Lyte, Slow Infusion; Saline 0.9%, Slow Infusion
Other: Fast Infusion Speed — Whenever fluid expansion is deemed necessary by the attending physician, infusion speed will be set at 999 mL/h. NOTE: This intervention will not be blinded.
  Arms: Plasma-Lyte, Fast Infusion; Saline 0.9%, Fast Infusion

SUMMARY:
A 2x2 factorial randomized study to evaluate the effect of a balanced crystalloid solution compared with 0.9% saline, and of rapid vs. slow infusion on clinical outcomes of critically ill patients

DETAILED DESCRIPTION:
Pragmatic, multicenter, 2x2 factorial randomized study. Severe patients admitted to the ICU at moderate to high risk for death or acute kidney injury will be randomly allocated to receive a balanced crystalloid solution (Plasma-Lyte®) or 0.9% saline and to receive crystalloids by rapid bolus infusion (999 mL/h) or slow infusion (333 mL/h) whenever plasma expansion is needed.

ELIGIBILITY:
Inclusion Criteria (all three):

1. Need for plasma expansion, and the clinician considers that Plasma-Lyte® or 0.9% saline are equally appropriate for patients, with no specific indications or contraindications for any of the fluids or for rapid or slow infusion.
2. Patients not expected to be discharged on the day after their admission.
3. At least one of the following risk factors for acute renal injury:

   1. Age ≥ 65 years
   2. Hypotension (mean arterial pressure [MAP] < 65 mmHg or systolic blood pressure [SBP] < 90 mmHg) or use of vasopressors
   3. Sepsis
   4. Use of invasive mechanical ventilation or of continuous noninvasive mechanical ventilation (including high-flow nasal cannula) > 12 hours
   5. Oliguria (< 0.5 mL/kg/hour for ≥ 3 hours)
   6. Serum creatinine ≥ 1.2 mg/dL for women or ≥ 1.4 mg/dL for men
   7. Liver cirrhosis or acute liver failure

Exclusion Criteria (any of the below):

1. Age < 18 years
2. Acute renal failure treated with renal replacement therapy (RRT) or expected to require RRT within the next 6 hours
3. Severe hyponatremia (serum sodium ≤ 120 mmol/L)
4. Severe hypernatremia (serum sodium ≥ 160 mmol/L)
5. Death considered imminent and inevitable within 24 hours
6. Patients with suspected or confirmed brain death
7. Patients under exclusive palliative care
8. Patients previously enrolled in the BaSICS study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11075 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days

SECONDARY OUTCOMES:
Renal failure requiring renal replacement therapy | 90 days
Renal Injury (KDIGO equal or greater than 2) | Days 3 and 7
Hepatic, cardiac, neurological, coagulation, and respiratory dysfunctions (assessed by Sequential Organ Failure Assessment [SOFA] scores) | Days 3 and 7
Mechanical ventilation free days | 28 days

OTHER OUTCOMES:
Intensive Care Unit Mortality | At ICU discharge, up to 90 days
Hospital Mortality | At Hospital discharge, up to 90 days
Length of Intensive Care Unit stay | At ICU discharge, up to 90 days
Length of hospital stay | At hospital discharge, up to 90 days
Quality of Life at 6 months | 180 days
  Assessed using EQ-5D. Will only be performed in a subsample of all included patients (10%)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre B Cavalcanti, MD, PhD, Study Chair — Hospital do Coracao; Fernando G Zampieri, MD, Principal Investigator — Hospital do Coracao; Nilton Brandao, MD, PhD, Study Director — Hospital Moinhos de Vento; Flávia R Machado, MD, PhD, Study Director — Universidade Federal de São Paulo, UNIFESP; Rodrigo S Biondi, MD, Study Director — Instituto de Cardiologia do Distrito Federal, ICDF; Flávio G Rezende de Freitas, MD, PhD, Study Director — Universidade Federal de São Paulo, Departamento de Cirurgia
Locations (1):
- Alexandre Biasi Cavalcanti, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be publicly available two years after trial results have been published

REFERENCES:
- [Derived] Zampieri FG, Damiani LP, Biondi RS, Freitas FGR, Veiga VC, Figueiredo RC, Serpa-Neto A, Manoel ALO, Miranda TA, Correa TD, Azevedo LCP, Silva NBD, Machado FR, Cavalcanti AB; BRICNet. Effects of balanced solution on short-term outcomes in traumatic brain injury patients: a secondary analysis of the BaSICS randomized trial. Rev Bras Ter Intensiva. 2022 Oct-Dec;34(4):410-417. doi: 10.5935/0103-507X.20220261-pt. Epub 2023 Mar 3. PMID 36888820
- [Derived] Zampieri FG, Damiani LP, Bagshaw SM, Semler MW, Churpek M, Azevedo LCP, Figueiredo RC, Veiga VC, Biondi R, Freitas FR, Machado FR, Cavalcanti AB; BRICNet. Conditional Treatment Effect Analysis of Two Infusion Rates for Fluid Challenges in Critically Ill Patients: A Secondary Analysis of Balanced Solution versus Saline in Intensive Care Study (BaSICS) Trial. Ann Am Thorac Soc. 2023 Jun;20(6):872-879. doi: 10.1513/AnnalsATS.202211-946OC. PMID 36735931
- [Derived] Zampieri FG, Damiani LP, Biondi RS, Freitas FGR, Veiga VC, Figueiredo RC, Serpa-Neto A, Manoel ALO, Miranda TA, Correa TD, Azevedo LCP, Silva NB, Machado FR, Cavalcanti AB; BRICNet. Hierarchical endpoint analysis using win ratio in critical care: An exploration using the balanced solutions in intensive care study (BaSICS). J Crit Care. 2022 Oct;71:154113. doi: 10.1016/j.jcrc.2022.154113. Epub 2022 Jul 14. PMID 35843046
- [Derived] Zampieri FG, Machado FR, Biondi RS, Freitas FGR, Veiga VC, Figueiredo RC, Lovato WJ, Amendola CP, Serpa-Neto A, Paranhos JLR, Lucio EA, Oliveira-Junior LC, Lisboa TC, Lacerda FH, Maia IS, Grion CMC, Assuncao MSC, Manoel ALO, Correa TD, Guedes MAVA, Azevedo LCP, Miranda TA, Damiani LP, Brandao da Silva N, Cavalcanti AB. Association between Type of Fluid Received Prior to Enrollment, Type of Admission, and Effect of Balanced Crystalloid in Critically Ill Adults: A Secondary Exploratory Analysis of the BaSICS Clinical Trial. Am J Respir Crit Care Med. 2022 Jun 15;205(12):1419-1428. doi: 10.1164/rccm.202111-2484OC. PMID 35349397
- [Derived] Zampieri FG, Machado FR, Biondi RS, Freitas FGR, Veiga VC, Figueiredo RC, Lovato WJ, Amendola CP, Assuncao MSC, Serpa-Neto A, Paranhos JLR, Andrade J, Godoy MMG, Romano E, Dal Pizzol F, Silva EB, Silva MML, Machado MCV, Malbouisson LMS, Manoel ALO, Thompson MM, Figueiredo LM, Soares RM, Miranda TA, de Lima LM, Santucci EV, Correa TD, Azevedo LCP, Kellum JA, Damiani LP, Silva NB, Cavalcanti AB; BaSICS investigators and the BRICNet members. Effect of Slower vs Faster Intravenous Fluid Bolus Rates on Mortality in Critically Ill Patients: The BaSICS Randomized Clinical Trial. JAMA. 2021 Sep 7;326(9):830-838. doi: 10.1001/jama.2021.11444. PMID 34547081
- [Derived] Zampieri FG, Machado FR, Biondi RS, Freitas FGR, Veiga VC, Figueiredo RC, Lovato WJ, Amendola CP, Serpa-Neto A, Paranhos JLR, Guedes MAV, Lucio EA, Oliveira-Junior LC, Lisboa TC, Lacerda FH, Maia IS, Grion CMC, Assuncao MSC, Manoel ALO, Silva-Junior JM, Duarte P, Soares RM, Miranda TA, de Lima LM, Gurgel RM, Paisani DM, Correa TD, Azevedo LCP, Kellum JA, Damiani LP, Brandao da Silva N, Cavalcanti AB; BaSICS investigators and the BRICNet members. Effect of Intravenous Fluid Treatment With a Balanced Solution vs 0.9% Saline Solution on Mortality in Critically Ill Patients: The BaSICS Randomized Clinical Trial. JAMA. 2021 Aug 10;326(9):1-12. doi: 10.1001/jama.2021.11684. Online ahead of print. PMID 34375394
- [Derived] Zampieri FG, Azevedo LCP, Correa TD, Falavigna M, Machado FR, Assuncao MSC, Lobo SMA, Dourado LK, Berwanger O, Kellum JA, Brandao N, Cavalcanti AB; BaSICS Investigators and the BRICNet. Study protocol for the Balanced Solution versus Saline in Intensive Care Study (BaSICS): a factorial randomised trial. Crit Care Resusc. 2017 Jun;19(2):175-182. PMID 28651514